CLINICAL TRIAL: NCT04883424
Title: The Effect of Family Support on Diabetes Patients' Health Beliefs, Behavioral and Metabolic Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08 / 262-320
Record Dates: First submitted 2021-04-26; First posted 2021-05-12 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Family Members; Diabetes Mellitus
Keywords: Family support; Diabetics; Health belief model; Diabet training
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Education Program Based on Health Belief Model (Experimental): Experimental group After the diabetic patients were determined according to the research criteria, they were randomly divided into intervention and control groups. First, pre-tests were applied to diabetics and family members in the experimental group. Diabetes Education Program Based on Health Belief Model It will be administered in two sessions to people with diabetes and their family members. This program; definition of diabetes, the importance of healthy nutrition in diabetes, the importance of exercise, the importance of regular medication, fingertip blood glucose measurement, acute and chronic problems that may develop in diabetic patients, diabetic foot care, personal self-care and family support. A reminder text message will be sent twice a week to diabetics and family members in the intervention group to manage their diabetes well. Once a month, both the diabetic patient and their family member will be called by phone for counseling.
  Interventions: Behavioral: Diabetes Education Program Based on Health Belief Model
- Control Group (No Intervention): First of all, pre-tests will be applied to diabetic patients in the control group. Diabetics in this group will not be intervened and their final tests will be made 3 months after the pre-test.

INTERVENTIONS:
Behavioral: Diabetes Education Program Based on Health Belief Model — After the application, increase in family support and decrease in blood sugar levels are expected in diabetic patients. Family members' diabetic attitudes are expected to increase.
  Arms: Diabetes Education Program Based on Health Belief Model

SUMMARY:
This study, designed according to the randomized pre-test and post-test control group experimental model, will be carried out with the patients who apply to the Diabetes Education Unit of Samsun Training and Research Hospital The universe of the study will consist of adult patients between the ages of 20-65 among the diabetic patients who apply to Samsun Training and Research Hospital Diabetes Education Unit.

The sample of the study will consist of 100 diabetic patients who comply with the selection criteria and volunteer to participate in the study. The average scores of Hensarling's Diabetes Family Support Scale in Diabetes Patients were determined as 64.12, with an error margin of %5% and a 95% confidence interval, with a sample size of 80% with a sample size of 35 patients for each group, a total of 70 patients.

Considering the participant losses during the project, 50 diabetic patients (experiment = 50, control = 50) for each group were determined as a total sample group of 100 diabetic patients with 50% reserve. Personal questionnaire prepared by the researcher in line with the literature, Health Belief Model Scale in Diabetes Patients, Hensarling's Diabetes Family Support Scale and Diabetes Attitude Scale will be used. The purpose of the study will be explained to the diabetic patients who apply to Samsun Training and Research Hospital Diabetes Education Unit and the study will be carried out with diabetic patients who agree to participate in the study. Diabetes patients will be divided into experimental and control groups by Simple Random Method. A training program will be applied to the diabetic patient and their family members included in the experimental group. After the training, a reminder text message will be sent to their phones twice a week for three months and they will be called once a month. Three months after the end of the training, the control will be called for examination.

DETAILED DESCRIPTION:
This study focuses on the effect of family support on diabetes management by using the Health Belief Model. This work; The health belief model, which is a human behavioral model, will comprehensively examine the effects of the planned diabetes education to be given to the diabetic patient together with the family member on the diabetes management of the diabetic patient.

Study design and environment The study is an experimental study with randomized controlled pre-test and post-test control group. The randomized clinical trial is based on guidelines recommended by Consolidated Standard of Reporting Trials - CONSORT 2010. The data of the study will be collected in the Diabetes Education Unit of Samsun Training and Research Hospital between January and June 2021.

As a pre-test for diabetic patients who applied to Samsun Training and Research Hospital Diabetes Education Unit and accepted to participate in the study; The questionnaire form prepared by the researcher in accordance with the literature, the Health Belief Model Scale in Diabetes Patients and Hensarling's Diabetes Family Support Scale will be applied. After the pretest application, they will be randomly assigned to the sample pool to be divided into experimental and control groups. Diabetes patients will be divided into experimental and control groups by simple random method. A questionnaire form prepared by the researcher in accordance with the literature and the Diabetes Attitude Scale will be applied to the family members of the diabetes patients in the experimental group.

Data Collection Tools Personal Information Form (for diabetic patients): This form, developed by researchers in accordance with the literature, is used by diabetic patients; It includes information about the disease such as age, gender, marital status, educational status, occupation, income status, duration of diabetes, history of other chronic diseases, diabetes treatment, alcohol-smoking, physical activity, nutrition, diabetes control interval.

Personal Information Form (for family member): This form, developed by researchers in accordance with the literature, consists of introductory features of the family member including gender, age, marital status, educational status, occupation, income, employment status, and relationship with a diabetic patient.

Health Belief Model Scale in Diabetes Patients: This scale; It is the form of "Health Belief Model Scale in Diabetes" adapted to Type 2 diabetes patients by Tan in 2004 and adapted to Turkish in 2007 by Kartal and Özsoy. There are 5 sub-dimensions of the model in the scale.

In the evaluation of the scale, Likert type scoring with scale items ranging from 1 to 5; "Strongly disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "strongly agree" (5). The scale consists of 33 items and five main sub-dimensions: Perceived sensitivity (4 items), Perceived severity (3 items), Perceived usefulness (7 items), Perceived barriers (9 items), and recommended health-related activities (10 items). A minimum of 33 and a maximum of 165 points can be obtained from the whole scale.

Hensarling's Diabetes Family Support Scale: The scale was developed by Hensarling in 2009 as a valid and reliable test that measures the perceived family support of adults with Type 2 diabetes. Turkish validity and reliability were established in 2011 by Akin.

As a result of the analysis, it determined 4 sub-dimensions of "Diabetes Family Support": empathic support (9 items), encouragement (7 items), facilitative support (6 items), and sharing support (2 items).

Each question with a scale consisting of a total of 24 questions is evaluated over 5 options. These options are "Never", "Almost Never", "Sometimes", "Most of the time", "Always".

The lowest possible score for Hensarling's Diabetes Family Support Scale is zero (0), and the highest possible total score is ninetysix (96). The fact that the total score obtained from the scale is close to 96 points indicates high family support. The fact that the score obtained from the scale is close to 0 points indicates that family support is perceived less.

Diabetes Attitude Scale (DAS): The Diabetes Attitude Scale, which was developed by the United States National Diabetes Commission and whose validity and reliability study was conducted in 1999 by Özcan, will be used to determine the attitudes of the individuals participating in the study. Seven subgroups covered by the DAS; special education need, attitude towards patient compliance, severity of type 2 diabetes, blood glucose control and complications, the effect of diabetes on the patient's life, attitude towards patient autonomy and attitude towards team care.

The number of items in the subgroups ranges from 3 to 7. Scale items were scored with Likert type scoring ranging from 1 to 5. If the score is> 3, it indicates positive attitude, if the score is 3, it indicates negative attitude. The increase of the score towards 5 or the decrease towards 1 strengthens the attitude in that direction. By adding up all the item scores of each subgroup of the scale and dividing it by the number of subgroup items, the attitude score of that individual belonging to the subgroup, ranging from 1 to 5, is calculated. Likewise, the diabetes attitude score is calculated in general by adding the scores of all items in the scale and dividing them by 34. The interpretation of the scale total score is similar to the interpretation of item scores. If the scale score is> 3, it indicates positive attitude, if the scale score is 3, it indicates a negative attitude, and the increase or decrease in the score strengthens the attitude in that direction.

Metabolic Results Control Form: This form was developed by the researchers in line with the literature. Before the pre-tests, the fasting blood glucose (FBG), Hemoglobin A1C (HbA1C), body mass index (BMI), blood pressure measurement, waist circumference measurement, triglyceride, HDL (high density lipoprotein), LDL (low density lipoprotein) lipoprotein) and total cholesterol values will be recorded.

Behavior Evaluation Form: This form was developed by researchers in line with the literature. In the pre-test, it is a 11-question form that includes the practices of diabetic patients in the experimental and control groups for diabetes management such as physical activity, nutritional habits, blood glucose monitoring and foot care.

As a result of the research, the data obtained from the personal information form, health belief model scale in diabetes patients, Hensarling's diabetes family support scale, behavior evaluation form and metabolic results form will be evaluated and reported in the SPSS package program. Descriptive statistics, paired t test, correlation analysis will be used to evaluate the data.

Ethical issues: Study approval was given by the Ondokuz Mayıs University Clinical Research Ethics Committee. (Decision No: B.30.2.ODM.0.20.08 / 262-320). All participants were informed about this study and written informed consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Type 2 Diabetes in the last 6 months
* Living in Samsun
* Being between the ages of 20-70
* HbA1c ≥ 6.5%
* Understanding and speaking Turkish
* Owning a smartphone and communicating with the phone
* Having blood glucose measurement tools at home
* Volunteering to participate in study with a family member of their choice

Exclusion Criteria:

* Being pregnant
* Having advanced or terminal disease (such as cancer, chronic kidney failure)
* Using an insulin pump
* Being disabled

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Health Belief Model Scale in Diabetes Patients | 3 months
  Health Belief Model Scale in Diabetes Patients: This scale; It is the "Health Belief Model Scale in Diabetes" form adapted by Tan in 2004 for Type 2 diabetes patients and adapted into Turkish in 2007 by Kartal and Ozsoy. The model in the scale has 5 sub-dimensions.
  In the evaluation of the scale, Likert type scoring with scale items between 1 and 5; "Strongly disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "strongly agree" (5). The scale consists of 33 items and five main sub-dimensions: perceived sensitivity (4 items), perceived severity (3 items), perceived usefulness (7 items), perceived barriers (9 items), and recommended health-related activities (10 items). A minimum of 33 and a maximum of 165 points can be obtained on the scale.
  In the posttest, it is aimed to increase the scale score in perceived sensitivity, perceived seriousness, perceived benefit and recommended activities related to health, and decrease the perceived barriers score.
Hensarling's Diabetes Family Support Scale | 3 months
  This scale determined 4 sub-dimensions of "Diabetes Family Support": empathic support (9 items), encouragement (7 items), facilitative support (6 items) and sharing support (2 items). A total of 24 questions are evaluated over 5 options. These options are "Never", "Almost Never", "Sometimes", "Most of the time", "Always". The lowest possible score for Hensarling's Diabetes Family Support Scale is zero (0) and the highest possible total score: ninetysix (96). The closer the Hensarling's Diabetes Family Support Scale total score is to the highest possible score of 96, the individual's perceived family support is expected. The closer the Hensarling's Diabetes Family Support Scale total score is to 0, the less family support is perceived.
  In the posttests, it is aimed to increase the score obtained from this scale.
HbA1c | 3 months
  HbA1c values of diabetic patients will be recorded before pre-tests. For these measurements, the latest examinations made in the hospital will be used. It is expected that the HbA1c values of diabetic patients will decrease in the posttest at the end of the third month.
Fasting Blood Glucose | 3 months
  Before the pre-tests, the fasting blood glucose value of diabetic patients will be recorded. For these measurements, the latest examinations made in the hospital will be used. It is expected that the HbA1c values of diabetic patients will decrease in the posttest at the end of the third month.
Diabetes Attitude Scale | 3 months
  The seven subgroups covered by the scale are special education needs, attitude towards patient compliance, severity of type 2 diabetes, blood glucose control and complications, the effect of diabetes on the patient's life, attitude towards patient autonomy and attitude towards team care. Scale items were scored with Likert type scoring ranging from 1 to 5. Score> 3 indicates positive attitude, score 3 indicates negative attitude. Increasing the score to 5 or decreasing to 1 strengthens the attitude in that direction.
  In the posttests, it is aimed to increase the diabetes attitude scale scores of family members in a positive way.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur AYDIN AVCI, Prof, Study Director — Ondokuz Mayıs University; Mustafa Kürşat ŞAHİN, Assoc.Prof, Study Chair — Ondokuz Mayıs University; Birsen ALTAY, Assoc.Prof, Study Chair — Ondokuz Mayıs University
Locations (1):
- Samsun Training and Research Hospital, Samsun, Turkey (Türkiye)